CLINICAL TRIAL: NCT02890316
Title: Cognitive and Emotional Assessment of Fatigue During Radiotherapy for Breast Cancer With and Without Homeopathy Treatment
Brief Title: Assessment of Fatigue During Radiotherapy for Breast Cancer With and Without Homeopathy Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Technion, Israel Institute of Technology (Other)
Responsible Party: Principal Investigator, Dr. Merav Ben-David, Head, Breast Radiation Unit, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2370-15
Record Dates: First submitted 2016-07-19; First posted 2016-09-07 (Estimated); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Radiation therapy with Homeopathy (Experimental): Patients in this arm will receive the homeopathy remedy during the adjuvant radiation therapy period, from treatment number 16 until the last assessment, 3 times every day.
  Interventions: Other: Homeopathy remedy; Radiation: Radiation as adjuvant therapy for breast cancer
- Radiation therapy with placebo (Placebo Comparator): Patients in this arm will receive the placebo remedy during the adjuvant radiation period, from treatment number 16 until the last assessment, 3 times every day.
  Interventions: Radiation: Radiation as adjuvant therapy for breast cancer

INTERVENTIONS:
Other: Homeopathy remedy — Homeopathy remedy, prescribed by a physician and prepared by licensed pharmacy.
  Arms: Radiation therapy with Homeopathy
Radiation: Radiation as adjuvant therapy for breast cancer — Daily radiation therapy.

SUMMARY:
To evaluate the effects of homeopathy treatment on radiotherapy-induced fatigue, cognitive and emotional functions.

DETAILED DESCRIPTION:
Sixty four female patients who underwent Chemotherapy and are planned to receive adjuvant whole breast radiation in the radiation departmental at the Sheba Medical Center, and who give a written consent for participation, will be included in the study.

Patients will undergo routine CT simulation and will receive 50 Gy in daily fractions of 2 Gy, five times a week (for total of 33 sessions during ~7 weeks, including boost of 8 fractions to the tumor bed) to the whole breast and lymphatic basins, according to the standard departmental protocol. Demographic and cancer treatment information will be collected, as well as Body mass index (BMI). At the first RT session (first assessment) and following 16-20 sessions of radiotherapy (second assessment), all patients will be evaluated for:

(i) fatigue level utilizing the Fatigue Symptom Inventory (FSI). (ii) attention performance utilizing the Pre-Pulse Inhibition (PPI) task. (iii) anxiety level utilizing both the startle response test and examining the Galvanic Skin Response (GSR) differences.

All examination will be conducted after the daily radiotherapy session. The homeopathic doctor will conduct an individual homeopathic evaluation during the second assessment meeting to all participants. According to these assessments, the pharmacist will prepare and provide 64 blinded numbered sets, 40 of which will contain the study remedy and 24 will contain the carrier only (i.e placebo).

Upon entry to the study after meeting the exclusion/inclusion criteria, a number from 1-64 will be drawn and the patient will receive the corresponding treatment.

The preparation of the homeopathic treatment (sugar globule containing the homeopathic dilution) is held in a licensed pharmacy and according to the Israeli Ministry of Health instructions of preparation. Sixty globules of sugar are wetted in the final diluted solution and dried for several minutes, and will be packed in the pharmacy to be consumed by the patients 3 times a day, 15 minutes before meal.

Placebo treatment is 1% sugar globule, similar in form and hedonic value of the aforementioned homeopathic globule.

During the 32-33 sessions of radiotherapy (third assessment), all patients will be re-assessed for the third time as before (i.e. first and second assessments). A fourth assessment to be held one month after the completion of radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged at least 18 years with unilateral breast cancer following chemotherapy.
2. Planned to receive 50 Gy whole breast irradiation and lymphatic basin + boost to tumor bed.
3. Capable of giving written informed consent following the instructions of receiving the study remedy or placebo.
4. No co-morbidities known to affect radiotherapy reactions.
5. No co-existing neurological or active psychiatric chronic diseases.
6. No evidence of infection or inflammation of breast to be treated.
7. Not receiving chemotherapy during radiotherapy course. Biological or hormonal therapy will be allowed during the study.

Exclusion Criteria:

1. Uncontrolled hypertension.
2. Participating in another clinical study with active treatment
3. Substance abuse.
4. Intellectual disabilities.
5. Unable to sign informed concent

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2016-07; Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Physiological monitoring of changes in anxiety during radiotherapy with and without homeopathy treatment. | Days 1, 16, 33 of radiation therapy
  Attention performance will be assessed by the Pre-Pulse Inhibition (PPI) task by evaluating the startle response test an Galvanic Skin Response differences.

SECONDARY OUTCOMES:
Physiological monitoring of changes in attention during radiotherapy with and without homeopathy treatment. | Days 1, 16, 33 of radiation therapy
  An interview assessing the changes attention with the Fatigue Symptom Inventory scale.

CONTACTS AND LOCATIONS:
Overall Officials: Merav Ben-David, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Merav Ben David, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dolev T, Ben-David M, Shahadi I, Freed Y, Zubedat S, Aga-Mizrachi S, Brand Z, Galper S, Jacobson G, Avital A. Attention Dysregulation in Breast Cancer Patients Following a Complementary Alternative Treatment Routine: A Double-Blind Randomized Trial. Integr Cancer Ther. 2021 Jan-Dec;20:15347354211019470. doi: 10.1177/15347354211019470. PMID 34027702